CLINICAL TRIAL: NCT07060027
Title: The Effect Of Single Versus Double Screws In Tenting Screw Technique For Horizontal Ridge Augmentation Before Dental Implant Placement (Randomized Clinical Trial)
Brief Title: Single vs. Double Tenting Screws for Horizontal Ridge Augmentation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omar Saad (Other)
Responsible Party: Sponsor-Investigator, Omar Saad, Principal Investigator - Teaching Assistant of Periodontology, Faculty of dentistry, Minia university, Minia University
Organization: Minia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4/626/88/2022
Record Dates: First submitted 2025-06-10; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Bone Defects

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Single tenting screw (Experimental): 8 patients indicated for lateral ridge augmentation in premolar-molar area (class I Seibert's classification) will be candidates to screw tent technique using single screw at crest position
  Interventions: Procedure: horizontal bone augmentation using single tenting screw
- Double tenting screw (Active Comparator): 8 patients indicated for lateral ridge augmentation in premolar-molar area (class I Seibert's classification) will be candidates to screw tent technique using double screws, one at a crestal position and the other one 5 mm apical to the first one.
  Interventions: Procedure: horizontal bone augmentation using Double tenting screw

INTERVENTIONS:
Procedure: horizontal bone augmentation using single tenting screw — Patients in this group will undergo guided bone regeneration (GBR) using a single titanium bone screw placed in the crestal position to stabilize the graft material. The surgical procedure includes sulcular and vertical releasing incisions, elevation of full-thickness buccal and palatal/lingual flaps, and multiple cortical perforations to enhance angiogenesis. The defect will be filled with particulate allograft extended 10-12 mm apicocoronally and covered with a bovine pericardium membrane. A tension-free primary closure will be achieved using 5-0 polypropylene sutures. Bone screw removal and implant placement will occur 6 months postoperatively. This group is distinguished by the use of a single crestal screw for graft stabilization compared to dual-screw fixation in the control group.
  Arms: Single tenting screw
Procedure: horizontal bone augmentation using Double tenting screw — Participants in this group will receive guided bone regeneration (GBR) with two titanium bone screws for enhanced graft stabilization. One screw will be placed at the crestal level, while a second screw will be inserted 5 mm apical to the first, providing vertical stabilization of the graft material. The procedure involves sulcular and vertical releasing incisions, full-thickness flap elevation on both buccal and palatal/lingual aspects, and multiple cortical perforations to stimulate vascularization. The defect will be filled with particulate allograft extending 10-12 mm apicocoronally and covered with a bovine pericardium membrane. Tension-free primary closure will be performed using 5-0 polypropylene sutures. At 6 months, screws will be removed and dental implants placed. This intervention is distinguished by the dual-screw fixation technique, designed to provide greater mechanical stability compared to the single-screw approach used in the comparator group.
  Arms: Double tenting screw

SUMMARY:
The goal of this clinical trial is to learn if using two screws works better than one screw for building up jawbone width before dental implant placement. It will also check the safety of both techniques. The main questions it aims to answer are:

* Does using two screws give better bone growth than using one screw?
* Which technique creates more stable bone for dental implants?

Researchers will compare the single-screw technique to the double-screw technique to see which works better for jawbone reconstruction.

Participants will:

* Receive either one or two small titanium screws placed in their jawbone to support a bone graft
* Have the graft covered with a protective membrane
* Return after 6 months for screw removal and dental implant placement
* Attend follow-up visits to check healing progress

The study will help dentists determine the best method for patients who need jawbone reconstruction before getting dental implants. All procedures use FDA-approved materials and follow standard surgical protocols.

New chat

ELIGIBILITY:
Inclusion Criteria:

* Patients are systemically healthy based on questionnaire dental modification of Cornell index (Bolender, C. L. et al., 1969).
* Gingival health according to the new classification system (Caton, J. G. et al., 2018).
* The recipient site of the augmentation is free from any pathological conditions.
* At least 1 tooth area with a ridge defect and planned to receive a dental implant. The site must be bordered by at least 1 tooth.
* Class I ridge defect according to Seibert's classification.
* Adequate interocclusal space to accommodate the available restorative components.

Exclusion Criteria:

* Parafunctional habits such as bruxism and clenching
* Smokers
* Pregnant females

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Change in Horizontal Ridge Width at Mid-Crestal Level | 6 months post-intervention
  Ridge width will be measured at the mid-crestal level using a bone caliper to the nearest millimeter. A standardized stent will ensure consistent measurement positioning.
Change in Horizontal Ridge Width 5 mm Apical to Crest | 6 months post-intervention
  Ridge width will be measured 5 mm apical to the crestal level using a bone caliper to the nearest millimeter. The same stent will standardize measurements.

SECONDARY OUTCOMES:
Change in Keratinized Mucosa Width at 6 Months Post-Reentry | 6 months post-intervention
  The width of keratinized mucosa will be measured using a periodontal probe to the nearest millimeter at the reentry procedure, 6 months after the initial intervention. The same stent will be used to standardize measurements.
Change in Alveolar Ridge Width via CBCT at 6 Months | 6 months post-intervention
  Cone-beam computed tomography (CBCT) will be used to assess changes in ridge width at 6 months post-intervention
Change in Bone Density via CBCT at 6 Months | 6 months post-intervention
  CBCT imaging will assess bone density changes (in Hounsfield units or grayscale values) at the treated site after 6 months.

CONTACTS AND LOCATIONS:
Locations (1):
- hospital of faculty of dentistry, Minia university, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT07060027/Prot_000.pdf